CLINICAL TRIAL: NCT06800339
Title: A Phase I, Single-Arm, Single-Institution Study Evaluating Neoadjuvant Chemoimmunotherapy With Immunosensitizing Radiation for Borderline Resectable Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating Neoadjuvant Chemoimmunotherapy With Immunosensitizing Radiation for Borderline Resectable Non-Small Cell Lung Cancer
Acronym: NEORADJUVANT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Matthew Ferris, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00112115
Record Dates: First submitted 2025-01-27; First posted 2025-01-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Radiation Treatment; SBRT; ChemoImmunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+Chemoimmunotherapy +/-Surgery (Experimental): Standard of care chemotherapy along with nivolumab. Nivolumab will be infused every 3 weeks for up to 3 cycles. Chemotherapy options include: carboplatin or cisplatin along with pemetrexed, paclitaxel or gemcitabine. Concurrently patient will receive 3 fractions of SBRT. Patient will then be evaluated for possible surgical resection.
  Interventions: Drug: Nivolumab; Drug: Chemotherapy; Radiation: SBRT; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Nivolumab — This will be administered intravenously once every 3 weeks for up to 3 cycles (i.e. 9 weeks of total systemic therapy)
Drug: Chemotherapy — Chemotherapy options include: carboplatin or cisplatin along with pemetrexed, paclitaxel or gemcitabine
Radiation: SBRT — Three fractions of radiation delivered every other day, for three total days. The final dose of radiation will happen within 7 days of starting chemoimmunotherapy
Procedure: Surgical Resection — Post treatment patient will be evaluated for surgical resection

SUMMARY:
The purpose of this research study is to find out if adding radiation prior to chemoimmunotherapy and surgery is effective for people with non-small cell lung cancer (NSCLC) who have the potential for surgery.

Standard of Care Chemoimmunotherapy:

For this study, standard of care chemotherapy will be used. This means this is the type of chemotherapy that is normal for your cancer. In addition to the chemotherapy, you will also receive the immunotherapy drug, nivolumab. This will be administered intravenously once every 3 weeks for up to 3 cycles (i.e. 9 weeks of total systemic therapy), prior to surgical resection assessment. This combination is made up of the chemotherapy drugs carboplatin or cisplatin along with pemetrexed, paclitaxel or gemcitabine, and the immunotherapy drug is nivolumab. The chemotherapy is used to kill cancer cells, and the immunotherapy enables your immune system to attack cancer cells.

Stereotactic Body Radiation Therapy (SBRT) SBRT is when radiation is delivered at higher doses over a smaller period of time. For this study, you will receive three doses of radiation delivered every other day, for three total days. The final dose of radiation will happen within 7 days of starting chemoimmunotherapy.

You will be followed for up to 100 days following your last chemoimmunotherapy dose to monitor for potential side effects. Following this you will continue with your standard follow up with your doctor. During the standard follow-up time, study staff will review your charts to see if there have been any new updates with your cancer following treatment so they can tell how this treatment affects how long patients live and whether it helps avoid recurrence of the cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to18 years at time of study entry
2. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
3. Participants with histologically confirmed stage II-IIIC(N3) NSCLC (per the 8th International Association for the Study of Lung Cancer) with disease that is considered borderline resectable prior to initiation of RT or systemic therapy.

   a. Patients with intrathoracic, contralateral N3 disease will be allowed to enroll (see exclusion criteria for further details)
4. Subject cases must be reviewed in a multidisciplinary thoracic tumor board setting prior to enrollment to allow for adequate discussion regarding the potential for resection.
5. Participants must have a tumor tissue sample available for biomarker testing, including next-generation sequencing to confirm EGFR/ALK status. Assessment of EGFR/ALK status may be performed locally through a CLIA approved laboratory testing method.

   a. Tissue source may be a formalin fixed paraffin block (FFPE) of a previous tumor biopsy sample. Source of biomarker testing may be obtained from archived tissue if adequate or from a new biopsy, if needed and clinically indicated
6. Absence of major associated pathologies that increase the surgery risk to an unacceptable level
7. Pulmonary function capacity (eg. FVC, FEV1, TLC, and DLCO) capable of tolerating proposed lung resection according to surgeon.
8. Adequate normal organ and marrow function defined below:

   1. Platelet count greater than or equal to100,000/mm3
   2. Hemoglobin greater than or equal to 8 g/dL
   3. Absolute neutrophil count (ANC) greater than or equal to 1000/mm3
   4. Creatinine less than or equal to 1.5 x ULN or creatinine clearance (CrCl) greater than or equal to 40 mL/min
   5. Total bilirubin less than or equal to 1.5 x ULN (except subjects with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL)
   6. AST, ALT, Alkaline phosphatase less than or equal to 3 x ULN per local testing
9. Subjects are deemed capable of giving informed consent and must have signed and dated an IRB approved written informed consent form. This written consent must be obtained before the performance of any protocol related procedures that are not part of normal standard of care.
10. Women of childbearing potential (WOCBP) must have negative serum or urine pregnancy testing within 30 days of study start.

Exclusion Criteria:

1. Presence of metastatic (Stage IV) disease, including malignancy pleural effusions.
2. Participants with N3 disease involving ipsilateral or contralateral scalene or supraclavicular lymph nodes. In the case of clinical suspicion for involvement of these lymph nodes, pathologic confirmation and biopsy may be pursued to determine final eligibility.
3. Participants with known sensitizing EGFR (L858R or Exon 19 deletion) mutations or ALK translocation. If testing is done, an FDA approved assay should be used and testing can be performed locally.
4. Participants with brain metastases are excluded from this study. All patients should have pre-study MRI brain or CT head with contrast to confirm the absence of intracranial disease, per standard of care staging procedures.
5. Participants with active autoimmune disease which would preclude immunotherapy. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of external trigger are permitted to enroll.
6. Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of autoimmune disease.
7. Participants with serious or uncontrolled medical disorders.
8. Participants with large-cell neuroendocrine carcinoma tumor histology.
9. Prior administration of chemotherapy or any other cancer therapy for early-stage NSCLC.
10. Prior therapy with an anti-PD-(L)1, anti-CTLA-4 antibody or any other antibody targeting t-cell co-regulatory pathways.
11. Participants with active hepatitis B (positive hepatitis B surface antigen) or hepatitis C virus (positive HCV RNA).

    1. Participants with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody and the absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to randomization. HBV carriers or those participants requiring antiviral therapy are not eligible to participate.
    2. Participants positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
12. Participants with poorly controlled or untreated human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS). All of the following criteria are required to define an HIV infection that is well controlled and therefore eligible for enrollment: undetectable viral RNA, CD4 count greater than or equal to 350, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications.
13. Active prior malignancy within the previous 3 years, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast.
14. History of allergy or hypersensitivity to nivolumab, or chemotherapy agents.
15. History of allogeneic organ transplantation.
16. Female patients who are pregnant or actively breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control methods from time of screening to 90 days after completion of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Tolerability of Adding Sub-ablative, Immunosensitizing, Radiotherapy to Standard of Care Neoadjuvant Chemoimmunotherapy | 20 weeks post initiation of neoadjuvant therapy
  Evaluate the tolerability of adding sub-ablative, immunosensitizing, radiotherapy to standard of care neoadjuvant chemoimmunotherapy prior to surgery for resectable NSCLC, measured by the rate of DLTs from time of neoadjuvant therapy initiation to start of definitive therapy (either surgery or chemoimmunotherapy initiation).

SECONDARY OUTCOMES:
Number of adverse events assessment by CTCAE v5.0 that are related to treatment | 20-22 weeks post initiation of neoadjuvant therapy
  Determine the safety of adding sub-ablative, immunosensitizing, radiotherapy to standard of care neoadjuvant chemoimmunotherapy prior to definitive resection for resectable NSCLC, measured by the frequency of drug related adverse events, including serious adverse events, occurring up to the initiation of definitive therapy (either surgery or chemoimmunotherapy initiation). Safety will be measured by the frequency of drug related adverse events, including serious adverse events (defined by CTCAE version 5), occurring up until the time of definitive therapy initiation (either surgery or chemoradiotherapy).
Pathologic Complete Response Rate (pCR) | 20-22 weeks post initiation of neoadjuvant therapy
  Estimate the rate of pathologic complete response after adding immunosensitizing radiotherapy to neoadjuvant chemoimmunotherapy prior to definitive resection. pCR is defined as lack of any viable tumor cells after complete evaluation in the resected lung cancer specimen and all sampled regional lymph nodes as determined by central pathology review and described by IASLC 2020 assessment criteria. The measure of interest is the proportion of resected patients with 0% residual viable tumor cells within all resected tissue as assessed by the central pathology review.
Major Pathologic Response Rate (MPR) | 20-22 weeks post initiation of neoadjuvant therapy
  Estimate the rate of major pathologic response after adding immunosensitizing radiotherapy to neoadjuvant chemoimmunotherapy prior to definitive resection. MPR is defined as ≤ 10% viable tumor cells in resected tumor after complete evaluation in the resected lung cancer specimen as determined by central pathology review and described by IASLC 2020 assessment criteria. The measure of interest is the proportion of resected patients with ≤ 10% residual viable tumor cells within all resected tissue as assessed by the central pathology review.
Measure rate of definitive resection | 1 year post completion of accrual
  Establish the rate of definitive resection for patients with borderline resectable NSCLC treated with subablative radiotherapy followed by neoadjuvant chemoimmunotherapy.
  Rate of definitive resection will be measured as the percentage of participants who undergo a complete R0 resection of their disease after receiving neoadjuvant subablative radiotherapy followed by chemoimmunotherapy out of all treated participants.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Upper Chesapeake- Kaufman Cancer Center, Bel Air, Maryland
  - Baltimore Washington Medical Center- Tate Cancer Center, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No